CLINICAL TRIAL: NCT04513886
Title: Healing After Connective Tissue Graft Harvesting in the Palatal Area With and Without Suture: A Randomized Controlled Trial
Brief Title: Healing After Connective Tissue Graft Harvesting in the Palatal Area With and Without Suture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mariel Viviana Gómez (Other)
Collaborators: Maimonides University (Other)
Responsible Party: Sponsor-Investigator, Mariel Viviana Gómez, Associate Professor. Department of Postgraduate Periodontics., Maimonides University
Organization: Maimonides University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2310/18
Record Dates: First submitted 2020-08-10; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Wound Healing
Keywords: wound healing; palate; connective tissue harvesting; single incision

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of two groups in parallel for the duration of the study: This study was a non-masked, randomized, controlled clinical trial, with a parallel design, comparing early healing of palatal wounds after harvesting subepithelial connective tissue graft using the single incision technique, with and without palatal sutures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suture Group (Active Comparator): After harvesting a subepithelial connective tissue graft using the single incision technique collagen haemostatic sponge placement and subsequent compression with gauze soaked in saline for 5 minutes, a cross- mattress suture and interrupted single sutures were performed using nylon 5-0 when appropriate.
  Interventions: Procedure: Subepithelial connective tissue graft (SCTG) using the single incision technique, with and without suturing the palate
- no Suture Group (Experimental): After harvesting a subepithelial connective tissue graft using the single incision technique, collagen haemostatic sponge placement and subsequent compression with gauze soaked in saline for 5 minutes no suture was performed.
  Interventions: Procedure: Subepithelial connective tissue graft (SCTG) using the single incision technique, with and without suturing the palate

INTERVENTIONS:
Procedure: Subepithelial connective tissue graft (SCTG) using the single incision technique, with and without suturing the palate — A SCTG was harvested using the single incision technique described by Hürzeler & Weng. The palatal incisions were standardized to extend between the area between mesial of the canine and mesial of the first molar.In the Suture Group sites a cross- mattress suture and interrupted single sutures were performed using nylon 5-0 when appropriate. In the no Suture Group sites, no suture was performed. In both groups, a CHS was placed after removing the graft to achieve the haemostasis of the palate and subsequent compressed with gauze soaked in saline for 5 minutes.

SUMMARY:
This study evaluated the outcomes in the early healing of palatal wounds after harvesting a subepithelial connective tissue graft (SCTG) using the single incision technique with placement of a collagen haemostatic sponge (CHS) without suturing the palate. The primary outcome of this study was to evaluate the early wound healing index (EHI).

DETAILED DESCRIPTION:
The aim of this study was to compare the outcomes in the early wound healing after harvesting a subepithelial connective tissue graft (SCTG) using the single incision technique and collagen haemostatic sponge (CHS) placement, with and without suturing the palate. 36 subjects were randomized to receive (n=18, Suture group-SG) or not a suture (n=18, no Suture group-nSG). Outcomes variables were: Early healing index (EHI) at 7, 14 and 30 days, self-reported pain using a visual analogue scale (VAS) at 7 and 14 days, immediate (iB) and delayed bleeding (dB). Data obtained were compared by Fisher's exact test, T test for independent sample, Mann-Whitney test (U test) and Wilcoxon sign test as appropriate. The level of significance was set at p < 0.05. Statistical analysis was performed with Infostat version 2015.

ELIGIBILITY:
Inclusion Criteria

* Subjects with an indication of mucogingival surgery for single gingival recession treatment that required harvesting a subepithelial connective tissue graft
* Age >18 years ≤ 60 years.
* Periodontally and systemically healthy.
* Palatal fibromucosa width ≥ 2mm evaluated with a North Carolina probe placed perpendicular to the hard palate, prior to surgery.

Exclusion Criteria

* Smoking.
* Contraindications for periodontal surgery.
* Subjects presenting coagulation disorders (history of Haemophilia, von Willebrand disease or anticoagulant therapy).
* Subjects taking medications known to interfere with periodontal tissue health or healing.
* Subjects that had been operated on the palate (connective tissue removed) previously from that same donor area.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
Early healing index | Day 7 post surgery
  1. Complete flap closure without fibrin line at the palate; 2. Complete flap closure with fibrin line at the palate; 3. Complete flap closure with small fibrin clot(s) at the palate; 4. Incomplete flap closure with partial necrosis of the palatal tissue; 5. Incomplete flap closure with complete necrosis of the palatal tissue.
Early healing index | Day 14 post surgery
  1. Complete flap closure without fibrin line at the palate; 2. Complete flap closure with fibrin line at the palate; 3. Complete flap closure with small fibrin clot(s) at the palate; 4. Incomplete flap closure with partial necrosis of the palatal tissue; 5. Incomplete flap closure with complete necrosis of the palatal tissue.
Early healing index | Day 30 post surgery
  1. Complete flap closure without fibrin line at the palate; 2. Complete flap closure with fibrin line at the palate; 3. Complete flap closure with small fibrin clot(s) at the palate; 4. Incomplete flap closure with partial necrosis of the palatal tissue; 5. Incomplete flap closure with complete necrosis of the palatal tissue.

SECONDARY OUTCOMES:
Number of participants with immediate bleeding | immediately postsurgery
  An embedded gauze with saline was pressed on the palate wound for 5 minutes in both groups. Positive iB was recorded if once the gauze was removed, bleeding persisted. Compression was repeated as many times as necessary until bleeding was arrested. If this maneuver was not enough, additional actions should be performed to stop bleeding and the patient would be excluded from the study.
Number of participants with delayed bleeding | 7 days post surgery
  Any type of bleeding from the palatal area reported during the postoperative period was recorded as positive
Pain level / discomfort | first week after surgery,
  Pain level / discomfort experienced at the surgical site of the palate, was self-reported by the subject and registered with a Visual Analogue Scale (VAS). It was required to the subject to graduate their sensitivity using a scale of 10 cm marked in mm between 0 and 100, labelled numerically from 0 to 10. Zero corresponds to "no discomfort" and 10 "unbearable pain". All other possible adverse effects were also recorded.
Pain level / discomfort | second week after surgery,
  Pain level / discomfort experienced at the surgical site of the palate, was self-reported by the subject and registered with a Visual Analogue Scale (VAS). It was required to the subject to graduate their sensitivity using a scale of 10 cm marked in mm between 0 and 100, labelled numerically from 0 to 10. Zero corresponds to "no discomfort" and 10 "unbearable pain". All other possible adverse effects were also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mariel V Gómez, Assoc Prof, Study Director — Maimonides University; Guillermo Schinini, Assoc Prof, Principal Investigator — Maimonides University; Hugo J Romanelli, Chair Prof, Study Chair — Maimonides University; Diego Sales, Assist Prof, Principal Investigator — Maimonides University; Leandro Chambrone, Chair Prof, Principal Investigator — Ibirapuera University
Locations (1):
- Maimonides University, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maino GNE, Valles C, Santos A, Pascual A, Esquinas C, Nart J. Influence of suturing technique on wound healing and patient morbidity after connective tissue harvesting. A randomized clinical trial. J Clin Periodontol. 2018 Aug;45(8):977-985. doi: 10.1111/jcpe.12960. Epub 2018 Jul 24. PMID 29908088
- [Background] Stavropoulou C, Atout RN, Brownlee M, Schroth RJ, Kelekis-Cholakis A. A randomized clinical trial of cyanoacrylate tissue adhesives in donor site of connective tissue grafts. J Periodontol. 2019 Jun;90(6):608-615. doi: 10.1002/JPER.18-0475. Epub 2018 Dec 26. PMID 30517975
- [Background] Lorenzana ER, Allen EP. The single-incision palatal harvest technique: a strategy for esthetics and patient comfort. Int J Periodontics Restorative Dent. 2000 Jun;20(3):297-305. PMID 11203571
- [Background] Fickl S, Fischer KR, Jockel-Schneider Y, Stappert CF, Schlagenhauf U, Kebschull M. Early wound healing and patient morbidity after single-incision vs. trap-door graft harvesting from the palate--a clinical study. Clin Oral Investig. 2014 Dec;18(9):2213-9. doi: 10.1007/s00784-014-1204-7. Epub 2014 Feb 23. PMID 24562700
- [Background] Lektemur Alpan A, Torumtay Cin G. PRF improves wound healing and postoperative discomfort after harvesting subepithelial connective tissue graft from palate: a randomized controlled trial. Clin Oral Investig. 2020 Jan;24(1):425-436. doi: 10.1007/s00784-019-02934-9. Epub 2019 May 18. PMID 31104113
- [Background] Rossmann JA, Rees TD. A comparative evaluation of hemostatic agents in the management of soft tissue graft donor site bleeding. J Periodontol. 1999 Nov;70(11):1369-75. doi: 10.1902/jop.1999.70.11.1369. PMID 10588501
- [Background] Wessel JR, Tatakis DN. Patient outcomes following subepithelial connective tissue graft and free gingival graft procedures. J Periodontol. 2008 Mar;79(3):425-30. doi: 10.1902/jop.2008.070325. PMID 18315424
- [Background] Del Pizzo M, Modica F, Bethaz N, Priotto P, Romagnoli R. The connective tissue graft: a comparative clinical evaluation of wound healing at the palatal donor site. A preliminary study. J Clin Periodontol. 2002 Sep;29(9):848-54. doi: 10.1034/j.1600-051x.2002.290910.x. PMID 12423299
- [Result] Hurzeler MB, Weng D. A single-incision technique to harvest subepithelial connective tissue grafts from the palate. Int J Periodontics Restorative Dent. 1999 Jun;19(3):279-87. PMID 10635174